CLINICAL TRIAL: NCT07325552
Title: iStent Inject Versus Goniotomy With Kahook Dual Blade in Patients With Ocular Hypertension and Glaucoma
Brief Title: iStent Inject Versus Goniotomy With Kahook Dual Blade in Glauocma Treatment
Acronym: iSKDB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1779
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Open Angle Glaucoma (OAG)
Keywords: glaucoma; iStent inject; Kahook Dual Blade goniotomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Procedure: KDB (Active Comparator): Cataract surgery combined with Kahook Dual Blade goniotomy.
  Interventions: Device: Goniotomy with KDB blade goniotomy
- Procedure: iStent (Active Comparator): Cataract surgery in combination with iStent Inject W implantation
  Interventions: Device: Two iStent inject implanation

INTERVENTIONS:
Device: Goniotomy with KDB blade goniotomy — Goniotomy with KDB glide will be performed at the end of Cataract Surgery through the temporal cataract incision.
  Arms: Procedure: KDB
Device: Two iStent inject implanation — The two stents will be injected in Schlemms canal at the end of cataract surgery through the temporal cataract incision.
  Arms: Procedure: iStent

SUMMARY:
The purpose of the study is to investigate the efficacy of cataract surgery in combination with Kahook Dual Blade Glide goniotomy (KDB) or iStent Inject W Trabecular Microbypass Stent (Istent) in eyes with Open-angle glaucoma.

DETAILED DESCRIPTION:
Glaucoma patients with significant cataract are being informed about the study and potential risks, all participants giving written informed consent and meeting the criteria will become eligibility for study entry. Participants meeting the eligible requirements will be randomized to Cataract Surgery combined with Kahook Dual Blade Glide (50 patients) or iStent Inject W (50 patients).

ELIGIBILITY:
Inclusion Criteria:

* Only one eye per participant
* Clinically significant cataract
* Glaucoma or intraocular hypertension treated with one to four medications and no need for filtering glaucoma surgery at the time of study enrollment.
* Open chamber angle with Schaffer grading three to four in at least two quadrants

Exclusion Criteria:

* Previous glaucoma surgery, including cyclodestructive procedures.
* Selective Laser Trabeculoplasty (SLT) within 90 days prior to planned surgery.
* Exudative age-related macular degeneration, proliferative diabetic retinopathy, clinically significant corneal dystrophy, other eye disease that affect intraocular eye pressure or visual field.
* Unable to participate and make written consent due to another medical condition.

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of intraocular pressure lowering medications compared to baseline | From enrollment to the end of treatment at 12 months
  Accountability of intraocular pressure lowering medications used by the patient
Intraocular pressure measured by Goldmann applanation tonometry (GAT) | From enrollment to the end of treatment at 12 months
  Number of participants with ≥20 percent intraocular pressure reduction or reduction with ≥1 medication compared to baseline

SECONDARY OUTCOMES:
Number of participants with intraocular pressure ≤21 mm Hg, ≤18 mm Hg, ≤15 mm Hg and ≤12mm Hg | From enrollment to the end of treatment at 12 months
  Intraocular pressure measured by Goldmann applanation tonometry (GAT) at 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Medical University of Bialystok, Bialystok, Polska
  - Ophthalmology Clinic Medical University of Bialystok, Bialystok